CLINICAL TRIAL: NCT00414479
Title: Assessment of Anaemia Attributable to Schistosomiasis in School Children in Kenya: Mechanisms and Effect of Treatment
Status: Completed | Type: Observational
Sponsor: DBL -Institute for Health Research and Development (Other)
Other Study IDs: SRP-KY-DK-06
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Anaemia; Schistosomiasis Infection; Malaria; Iron Deficiency
Keywords: schistosomiasis; anaemia; malaria; iron deficiency
MeSH Terms: conditions — Anemia; Malaria; Iron Deficiencies; Schistosomiasis | interventions — Iron

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- children 9-12 years of age: Children with schistosomiasis, malaria and anaemia
  Interventions: Drug: praziquantl, iron, ACT

INTERVENTIONS:
Drug: praziquantl, iron, ACT

SUMMARY:
The purpose of this study is to determine the extend and the nature of anemia in school children and the correlation between anemia and schistosomiasis infections, malaria infections and/or malnutrition (iron deficiency).

DETAILED DESCRIPTION:
The study will be carried out in an area around Lake Victoria in Kenya where the prevalence of schistosomiasis and malaria are highest in the areas nearest to the Lake. Depending on the prevalence of schistosomiasis a sample of between 876 to 2.524 children will be enrolled in the study. The children who will be in the age between 9 to 12 year, will have their stool and urine examined for schistosomiasis and intestinal worms and a blood sample will be examined for malaria parasites and the hemoglobin level. Children will also be weight, measured and examined by a doctor and register their food intake over one week, to determine their nutritional status. Children who are found to be infected with schistosomiasis, intestinal worms or malaria will be offered treatment. Children who are found to have anemia will be offered a course of iron supplementation, children with severe anemia will be referred to the nearest health facility for treatment. 12 months after the initial examinations and treatment all children will have a re-examination of their stool, urine and blood.

ELIGIBILITY:
Inclusion Criteria:

* school children between 9 to 12 year

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children 9-12 years of age
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2006-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
hemoglobin level

SECONDARY OUTCOMES:
Schistosomiasis infection
malaria infection
iron deficiency

CONTACTS AND LOCATIONS:
Overall Officials: Diana Karanja, DR, Principal Investigator — Kenya Medical Research Institute
Locations (1):
- Kenya Medical Research Institute, Kisumu, Kenya